CLINICAL TRIAL: NCT06063772
Title: Effect of Treatment of Pre-induction Hypertension on Hemodynamic Stability During Induction of General Anesthesia
Acronym: INGRESS
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Edward O'Brien, Clinical Professor, Anesthesiology, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 807353
Record Dates: First submitted 2023-05-08; First posted 2023-10-03 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — clevidipine; Ringer's Lactate

STUDY DESIGN:
Intervention Model Description: Prospective blinded trial comparing the effect on post induction hemodynamic stability of pre-induction treatment of hypertension to placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: 1. Initial identification of patients will be based on measured blood pressure. No other criteria will be used to identify patients for screening.
  2. Cohort assignment will be made using a block randomization table.
  3. The investigator measuring hemodynamics in the OR during induction will be blind to the patient's cohort assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Clevidipine (Experimental): Once consented, patients will be randomized into one of two groups using a block randomization table. The treatment arm will receive clevidipine. Clevidipine comes from the manufacturer in a "ready to use" formulation. It requires no preparation by pharmacy, nursing or physician staff. All patients randomized to receive clevidipine will be in the experimental cohort.
  Interventions: Drug: Clevidipine
- Placebo (Lactated Ringers) (Placebo Comparator): The Control arm will receive Lactate Ringers as placebo. All patients randomized to receive lactated ringers will be in the control cohort. Lactated Ringers is stored at room temperature (25°C)
  Interventions: Drug: Lactated Ringers, Intravenous

INTERVENTIONS:
Drug: Clevidipine — The investigator will start the appropriate drug and titrate the drug in the pre-operative area until the mean arterial pressure is between 70 mmHg and 110 mmHg. The infusion will be titrated every 90 seconds to a maximum rate 32 mg/hr for clevidipine or the volume equivalent of placebo.
  Other Names: Cleviprex
  Arms: Clevidipine
Drug: Lactated Ringers, Intravenous — The investigator will start the appropriate drug and titrate the drug in the pre-operative area until the mean arterial pressure is between 70 mmHg and 110 mmHg. The infusion will be titrated every 90s to a maximum rate 32mg/hr for clevidipine or the volume equivalent of placebo.
  Other Names: Placebo
  Arms: Placebo (Lactated Ringers)

SUMMARY:
The purpose of this study is to determine if treatment of pre-induction hypertension with an intravenous short acting calcium channel antagonist will (1) reduce the magnitude and duration of blood pressure excursions outside of a pre-established normal range and (2) decrease the requirement for vasoactive medications during the period from induction of anesthesia until just prior to surgical incision.

DETAILED DESCRIPTION:
The investigators hypothesize that treatment of hypertension (defined as systolic blood pressure (SBP) > 140 mmHg or diastolic blood pressure (DBP) > 90 mmHg) with an IV short acting, calcium channel antagonist will (1) reduce excursions outside of a pre-specified blood pressure range and (2) reduce the requirement for exogenous vasopressor agents from the period of induction until incision in adults undergoing general anesthesia.

This is a single site, randomized, blinded, placebo controlled prospective trial during which the continuous intravenous administration of clevidipine or placebo will be administered to target a blood pressure in a specified normal range.

The trial will be performed by two investigators. The first investigator will work with the pre-operative nursing staff to identify patients in the pre-op waiting area who meet criteria for hypertension. Admission criteria to the study will be a systolic blood pressure in the Stage 2 category (between 140 mmHg and 180 mmHg or a diastolic blood pressure between 90 mmHg and 110 mmHg). These criteria are chosen based on the 2017 American Heart Association/American College of Cardiology guidelines where blood pressure greater than 180/110 mmHg is a hypertensive emergency and would prompt case cancellation and blood pressure < 140/90 mmHg would not require immediate pharmacological intervention.

Following an information session during which the consent document and the UCSD HIPPA form are reviewed, discussed and signed, participant will be assigned a study number and relevant baseline data will be collected from the patient's medical record including age, ASA classification, history of known cardiac, pulmonary, renal disease and home medications. Once consented, patients will be randomized into one of two groups using a block randomization table. The treatment arm will receive clevidipine and the control arm will receive a placebo solution (lactated Ringer's solution).

The investigator will start the appropriate drug and titrate the drug in the pre-operative area until the mean arterial pressure is between 70 mmHg and 110 mmHg. The infusion will be titrated every 90 seconds to a maximum rate 32 mg/hr for clevidipine (which is 64 ml/hr) or the volume equivalent of placebo. The investigator will measure the patient's vital signs every 3 minutes with initiation or change in infusion rate until the subject's mean arterial pressure is within the normal range and the subject is on a stable dose of the drug for two concurrent values. The dose will therefore be determined by the patient's response to the drug. This is not a dose-ranging or dose escalation study. After the blood pressure is stable, the investigator will measure and record the blood pressure every 15 minutes.

The patient will go to the OR with the drug or placebo infusing. A second investigator who is blinded to the identification of the drug will monitor the patient in the operating room. When the clinical anesthesia team is ready to induce anesthesia, the second investigator will stop the infusion and ask the clinicians to wait ninety seconds since clevidipine has a context-sensitive half-time of less than one minute, the plasma drug concentration will have declined by more than 87.5%. After ninety seconds, the clinicians will induce anesthesia for the patient with standardized doses of induction agents and standard vapor concentrations. The second investigator will record the blood pressure every minute in the operating room from the time of induction (administration of the first dose of sedative-hypnotic drug) until just prior to incision by the surgeon.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Any patient older than 18 years
4. Scheduled for elective surgery requiring general anesthesia
5. Presenting with hypertension during the pre-operative assessment (defined as either a systolic blood pressure > 140 mmHg or a diastolic blood pressure > 90 mmHg

Exclusion Criteria:

1. Known adverse reaction to clevidipine or any of its constituent parts.
2. Presence of structural heart disease.
3. Known acute or chronic kidney disease.
4. Pregnancy or lactation.
5. Non-elective surgery.
6. Treatment with another investigational drug or other intervention at the time of enrollment.
7. Patients unable to consent for themselves.
8. Incarcerated patients.
9. Known defect in lipid metabolism.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Magnitude and Duration of Deviation from a normal blood pressure range. | The investigators will measure and record blood pressure at 2 minute intervals from induction of anesthesia until just prior to incision.
  Blood pressure (systolic, diastolic and mean) will be recorded and plotted against time. The area under the curve of that plot that is outside of the normal blood pressure range is the outcome measure upon which the investigators will compare the clevidipine treated cohort to the placebo treated cohort.

SECONDARY OUTCOMES:
Dose of vasoactive drugs used during induction of anesthesia. | Investigators will record the dose of vasoactive drugs administered from induction until just prior to incision.
  All vasoactive drug name(s) and dose (s) will be recorded. The difference in doses will be compared between the clevidipine cohort and the placebo cohort.

CONTACTS AND LOCATIONS:
Overall Officials: Edward O O'Brien, M.D., Principal Investigator — University of California, San Diego

IPD SHARING:
Plan to Share IPD: No